CLINICAL TRIAL: NCT02313324
Title: The Effects of Extracorporeal Shock Wave Therapy in Patients With Coccydynia: A Randomized Controlled Trial
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kmutth-101-023
Record Dates: First submitted 2014-12-03; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2012-11

CONDITIONS: Coccydynia
Keywords: Coccydynia; Extracorporeal shock wave therapy; Disability
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESWT group (Experimental): The patients were randomly assigned to the extracorporeal shock wave therapy (ESWT) group.
  Interventions: Device: Extracorporeal shock wave therapy (ESWT)
- SWD combined IFC group (Active Comparator): The patients were randomly assigned to the SIT group. The patients received combined therapy with shortwave diathermy (SWD) and interferential current (IFC) performed by the same physiotherapist at each treatment session.
  Interventions: Device: SWD combined IFC

INTERVENTIONS:
Device: Extracorporeal shock wave therapy (ESWT) — The patients received 2000 shots of extracorporeal shock wave therapy in the coccyx area per session for four sessions (one session a week for 4 consecutive weeks). The frequency used was 5 Hz and the pressure was 3-4 bar.
  Arms: ESWT group
Device: SWD combined IFC — The shortwave diathermy (SWD) was the inductive mode with a coil at a frequency of approximately 27.12 MHz. The shortwave diathermy applicator was placed over the sacrococcygeal area. The treatment duration was 20 minutes. After completing the SWD treatments, the patients received the interferential current (IFC) treatment. IFC provides deeper electrical stimulation. The electrical current was applied to the gluteal area using four electrodes from 2 channels of the stimulator. The four electrodes were set on the gluteal area. The carrier frequency, typically 4000 Hz and 4100 Hz and designed to interfere with each other, resulted in a beat frequency of 100 Hz within the treated area. The treatment duration was 20 minutes. The protocol was set as 3 times per week for a period of 4 weeks.
  Arms: SWD combined IFC group

SUMMARY:
The purpose of this study is to evaluate the effects of extracorporeal shock wave therapy (ESWT) on the outcomes of coccydynia.

DETAILED DESCRIPTION:
Coccydynia is pain in the coccygeal region, and usually treated conservatively. Extracorporeal shock wave therapy (ESWT) was incorporated as non-invasive treatment of many musculoskeletal conditions. However, the effects of ESWT on coccydynia are less discussed. The purpose of this study is to evaluate the effects of ESWT on the outcomes of coccydynia. Patients were allocated to ESWT (n=20) or physical modality (SIT) group (n=21) randomly, and received total treatment duration of 4 weeks. The visual analog scale (VAS), Oswestry disability index (ODI), and self-reported satisfaction score were used to assess treatment effects. The VAS and ODI scores were significantly decreased after treatment in both groups, and the decrease in the VAS score was significantly greater in the ESWT group. The mean proportional changes in the ODI scores were greater in the ESWT group than in the SIT group, but the between-group difference was not statistically significant. The patients in the ESWT group had significantly higher subjective satisfaction scores than SIT group. The investigators concluded that ESWT is more effective and satisfactory in improving discomfort and disability caused by coccydynia than the use of physical modalities. Thus, ESWT is recommended as an optimal treatment option for patients with coccydynia.

ELIGIBILITY:
Inclusion Criteria:

* First-time diagnosed with coccydynia
* History of direct traumatic events to the buttocks, such as falls or slipping

Exclusion Criteria:

* Tumors of the cauda equina
* Pelvic surgery
* Herniation of the lumbosacral disc
* Internal procidentia
* Genitourinary or gastrointestinal complaints
* Psychogenic factors

Ages: 20 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from pre-enrollment in Visual analog scale (VAS) at 5th and 8th week after first intervention | pre-enrollment, 5th and 8th week after first intervention
  a scale from 0 through 100 (0 for no pain and 100 for the worst pain)

SECONDARY OUTCOMES:
Change from pre-enrollment in The Oswestry disability index (ODI, in Chinese) at 5th and 8th week after first intervention | pre-enrollment, 5th and 8th week after first intervention
  There are six statements to be ranked on a scale of 0 to 5 in each of the 10 sections of the questionnaire. The contents relate to impairments such as pain intensity and abilities in personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling. The patients were asked to identify the corresponding level of disability in each section. The total score ranges from 0 to 50; 0 represents the highest level of function, and 50 indicates completely disabled.
Change from pre-enrollment in Self-reported satisfaction scales at 8th week after first intervention | 8th week after first intervention
  A 5-level scale was used for evaluation at the 8th week after treatment. The excellent and good scores were categorized into one group, and the acceptable and poor scores were categorized into another group for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsin Chen, MD.PhD, Principal Investigator — Kaohsiung Municipal Ta-Tung Hospital

REFERENCES:
- [Derived] Lin SF, Chen YJ, Tu HP, Lee CL, Hsieh CL, Wu WL, Chen CH. The Effects of Extracorporeal Shock Wave Therapy in Patients with Coccydynia: A Randomized Controlled Trial. PLoS One. 2015 Nov 10;10(11):e0142475. doi: 10.1371/journal.pone.0142475. eCollection 2015. PMID 26556601